CLINICAL TRIAL: NCT07046858
Title: Predictive Accuracy of Platelet Lymphocyte Ratio & Platelet Neutrophil Ratio in Detecting Early Trauma Induced Coagulopathy
Brief Title: Predictive Accuracy of PLR and PNR in Detecting ETIC
Acronym: ETIC
Status: Recruiting | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Amrutha Thotten, Junior Resident, Jubilee Mission Medical College and Research Institute
Other Study IDs: 47/23/IEC/JMMC&RI
Record Dates: First submitted 2023-08-09; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Trauma Injury; Coagulopathy
Keywords: Early trauma induced coagulopathy
MeSH Terms: conditions — Accidental Injuries; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Trauma patients with and without ETIC: All the trauma patients coming to ED for whom the physician send investigations

SUMMARY:
Observational study to know what is the predictive accuracy of platelet-neutrophil ratio (PNR) and platelet-lymphocyte ratio (PLR) done in patients presenting to ED( emergency department)within 6 hours of trauma; in detecting early trauma induced coagulopathy during hospital admission

DETAILED DESCRIPTION:
Trauma has a significant impact on the wellbeing and healthcare for the populations. Millions of patients seek medical help as a result of trauma, with a substantial proportion of patients suffering from life-changing or life-limiting injuries. The leading cause of traumatic death worldwide is road traffic collision, followed by suicide and homicide.(4) The role of platelets in the hemostasis and coagulation is crucial. Platelet interaction with lymphocytes, neutrophils, and monocytes modifies both the innate and adaptive immune responses.Platelets stick to the damaged endothelium and recruit leukocytes to the sites of injury.

Lymphocytes are the major cellular components of the humoral and cell-mediated immune system which include T, B, and natural killer cells. Platelet-lymphocyte ratio (PLR), platelet- neutrophil ratio (PNR) could reflect the balance between the body response to inflammation and immunity mediators Previously, few studies have tested the usefulness of PLR, PNR for predicting the outcomes in stroke , cardiovascular diseases. abdominal trauma, ARDS (Acute Respiratory Distress Syndrome) & sepsis. I would like to do a study, where the results could be utilized in a resource limited hospital , for early referral and the prognostic value of these biomarkers in predicting ETIC in trauma.

The present study hypothesize that the on-admission PLR , PNR values would help early risk stratification and timely management of trauma patients which subsequently improve the outcomes

ELIGIBILITY:
Inclusion Criteria:

* All patients with trauma AND
* Presenting to ED within 6 hours of the event AND
* The ED Physician sends coagulation profile

Exclusion Criteria:

* Treated with intravenous fluids, drugs, whole blood and blood products elsewhere
* Patients admitted with a non-mechanical mechanism of injury, specifically drowning, hanging,or burns, as these mechanisms may result in a different biologic response than mechanical trauma
* Patients on known medications affecting coagulation profile or hemogram
* Patients with known chronic liver disease, chronic renal failure, malignancy, hematological disorders
* Patients not consenting for the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients with trauma AND Presenting to ED within 6 hrs of the event AND The ED Physician sends coagulation profile
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-10-27 (Estimated); Study Completion 2025-11-27 (Estimated)

PRIMARY OUTCOMES:
1. Sensitivity, specificity, positive and negative predictive value | 24 hours
  PLR and PNR ratio in predicting in-hospital transfusion requirement during index hospital admission.

SECONDARY OUTCOMES:
Compare the AUROC ( Area Under the Receiver Operating Characteristic Curve) of PLR and PNR ratio in predicting in-hospital transfusion requirement during index hospital admission | 24 hours
  PLR and PNR ratio in predicting in-hospital 30 day mortality
Compare the AUROC of PLR and PNR ratio in predicting prolonged ventilatory support (>21 days) | 24 hours
  Prolonged ventilators support
Compare the incidence of emergent surgery, renal replacement therapy amongst patients developing ETIC and those who do not during the duration of hospital stay or within 30 days (whichever is earlier) | 24hours
  Renal replacement therapy in patients with ETIC
Compare the length of hospital stay, total number of surgeries, total intensive care days in numbers amongst patients developing ETIC and those who do not during the duration of hospital stay or within 30 days (whichever is earlier) | 24hours
  length of hospital stay, total number of surgeries, total intensive care days in numbers amongst patients developing ETIC and those who do not during the duration of hospital stay or within 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Jubilee Mission Medical College, Thrissur, Kerala, India